CLINICAL TRIAL: NCT01512303
Title: Complementary and Alternative Interventions for Veterans With Posttraumatic Stress Disorder: Community Program Evaluation Study
Brief Title: Complementary and Alternative Interventions for Veterans With Posttraumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to funding issues
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: The Dana Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0641
Record Dates: First submitted 2012-01-06; First posted 2012-01-19 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: PTSD
Keywords: PTSD; Veterans' Health; Meditation; MRI, Functional
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Yoga; Mindfulness-Based Stress Reduction; Mindfulness; Meditation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sudarshan Kriya Yoga: SKY (Experimental): SKY incorporates yoga, discussion periods and several types of breathing exercises for relaxation. Initial breathing exercises are calming and focusing. Subsequent breathing exercises are more fully engaging energizing, allowing the practitioner to focus more fully in each moment. All are soothing and present-focused. Participants will be encouraged to learn all the breathing exercises, and to utilize the exercises the ones that seems most appropriate for their needs. 8-day intensive group class (2.5 hours/day) followed by 4 weekly sessions (3 hours/session).
  Interventions: Behavioral: Sudarshan Kriya Yoga
- Mindfulness-Based Stress Reduction: MBSR (Experimental): MBSR incorporates yoga, discussion periods, and several types of meditation, all involving attention to the present moment and acceptance of any feelings, sensations or thoughts, allowing the practitioner to calm his or her mind and come back to the present moment. The typical MBSR format will be adapted to match the SKY intervention. This intervention will include an 8-day intensive group class (2.5 hours/day) followed by 4 weekly sessions (3hrs/session).
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Wait-List Control: WLC (No Intervention): Participants will undergo no intervention. These participants will have the option of receiving one of the two interventions at the conclusion of the study.
- Non-PTSD control (No Intervention): Baseline measures only will be collected from a group of 50 combat-exposed veterans without PTSD to assess group differences on these measures prior to treatment.

INTERVENTIONS:
Behavioral: Sudarshan Kriya Yoga — SKY incorporates yoga, discussion periods and several types of breathing exercises for relaxation.
  Other Names: SKY; yoga
  Arms: Sudarshan Kriya Yoga: SKY
Behavioral: Mindfulness-Based Stress Reduction — MBSR incorporates yoga, discussion periods, and several types of meditation, all involving attention to the present moment and acceptance of any feelings, sensations or thoughts
  Other Names: MBSR; mindfulness; meditation
  Arms: Mindfulness-Based Stress Reduction: MBSR

SUMMARY:
The overarching aim of this proposal is to research whether meditation-based treatments are effective in decreasing posttraumatic stress disorder (PSTD) symptoms in veterans, which complementary and alternative (CA) treatments are most effective, and how individual differences predict treatment efficacy.

DETAILED DESCRIPTION:
The overarching purpose of this study is to assess the impact of CA interventions on posttraumatic stress symptoms in veterans with PTSD. Twenty percent of the approximately 2 million veterans returning from Iraq and Afghanistan ("Operation Iraqi Freedom" or OIF and "Operation Enduring Freedom" or OEF) suffer from the symptoms of Post-traumatic Stress Disorder. PTSD may be the reason behind alarming increases in suicidal behavior among returning veterans in Wisconsin and nation-wide. In addition to traditional treatments, Veterans Administration (VA) Hospitals and other community institutions for veterans now offer CA programs to their patients. Past research from our laboratory and others suggests that CA programs may provide effective relief from anxiety while increasing psychological well-being. However, little research exists on the effects of CA programs for combat veterans with PTSD. The proposed study aims to address this important gap by assessing CA programs such as Sudarshan Kriya Yoga (SKY) and Mindfulness-Based Stress Reduction (MBSR). 150 veterans with PTSD will be randomly assigned to either SKY, MBSR, or the wait-list control (WLC) group. We will assess participants' PTSD symptoms pre-intervention, post-intervention (approximately 10-14 days after initial visit), and 1 month post-treatment (approximately 6 weeks after initial visit). In order to evaluate the programs' effects as comprehensively as possible, we propose a multi-method approach: baseline psychophysiology, autonomic reactivity and recovery, neuropsychological (cognitive) assessments, self-report questionnaires, and functional brain imaging (fMRI). Baseline measures will be collected from a group of 50 combat-exposed veterans without PTSD to assess group differences on these measures prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* In the age range of 18-50.
* Capable of giving informed consent
* Fluent in English
* Exposure to one or more life-threatening war zone trauma events in Iraq or Afghanistan within the last 8 years.
* Pharmacological or psychotherapeutic treatment stable for at least 8 weeks prior to beginning of study
* Good general medical health (see Medical Exclusion Criteria)
* DSM-IV criteria for current PTSD as determined by CAPS (PTSD groups only)
* Combat-exposed, non-PTSD control veterans must be free of any current DSM-IV Axis I disorder
* Participants must agree to not begin a new course of treatment for the duration of the study

Exclusion Criteria:

* Weight of 352 pounds or over (due to constraints of MRI scanner)
* Women who are pregnant, planning to conceive during the research timeline, or breastfeeding will be excluded.
* Metallic implants such as prostheses or aneurysm clip, or electronic implants such as cardiac pacemakers
* Neurological or serious medical condition that may contraindicate MRI or that may overlap with physiological substrates of psychiatric conditions (see below for descriptions)
* History of seizures or seizure disorder
* Moderate or severe traumatic brain injury (over 30 minutes unconscious)
* Current active substance dependence or dependence within 3 months (other than nicotine)
* Meets DSM-IV criteria for bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorder NOS, delirium, or any DSM-IV cognitive disorder.
* Substance dependence disorder within 3 months or any current substance dependence
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior that poses an immediate danger to patient or others.
* Current use of benzodiazepines or beta-blockers
* Nonsuicidal depression comorbid with PTSD will NOT be exclusionary
* Extensive experience in yoga and meditation or have learned MBSR or SKY previously

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Clinician-Administered PTSD Scale (CAPS) scores | Baseline, 1 month post-intervention (approx. 6 weeks)
Change in PTSD Checklist-Military (PCL-M) scores | Baseline, Post-Intervention (approx. 10-14 days), 1 month post-intervention (approx. 6 weeks)
Change in fMRI brain blood oxygen level-dependent (BOLD) responses | Baseline, post-intervention (approx 10-14 days)
  Brain activation during anticipation of, response to, and recovery from aversive stimuli will be measured at baseline, and the intervention groups will be compared to the wait-list controls following the intervention to assess changes based on the interventions.

SECONDARY OUTCOMES:
Quality of sleep | Baseline through one month post-intervention (approx. 6 weeks)
  Sleep quality will be assessed using actigraphy
Changes in self-reported mood, anxiety, and sleep symptoms | Baseline, post-intervention (approx. 10-14 days), one month post-intervention (approx. 6 weeks)
Changes in peripheral psychophysiological arousal | Baseline and post-intervention (approx. 10-14 days)
  Assessed using multiple measures, including heart rate, heart rate variability, corrugator EMG, and skin conductance.
Changes in neuropsychological functioning | Baseline, post-intervention (approx. 10-14 days)
  Memory, attention, and rapid perceptual processing will be measured using neuropsychological tasks by Cambridge Cognition and/or the NIH toolbox

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Davidson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Waisman Center, University of Wisconsin, Madison, Wisconsin, United States